CLINICAL TRIAL: NCT03418870
Title: Improving Preterm Infant Outcomes With Family Integrated Care and Mobile Technology
Acronym: mFI-Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Los Angeles (Other); University of California, San Diego (Other); Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 16-19542
Record Dates: First submitted 2017-12-18; First posted 2018-02-01 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Premature Birth of Newborn
Keywords: Intensive Care Units, Neonatal; Parents; Mobile application
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Phase 1 is "usual care" and Phase 2 is the intervention phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Integrated Care (mFI-Care) (Experimental): Parents of infants assigned to the Family Integrated Care (mFI-Care) intervention will be treated as primary caregivers for their infants and participate in daily medical rounds, with mFI-Care-trained nurses serving as teachers and coaches. Parent training on the Canadian FI-Care Parent Curriculum will be provided during small group sessions facilitated by the study team. Parents will receive peer support from mFI-Care-trained alumni parents and can interact with other mFI-Care parents through the We3Health App secure online parent forum. mFI-Care parents will be expected to track time spent with their infant; record infant activity, feeds and output; track learning and skills acquisition; and keep a journal of the NICU experience using the We3Health app.
  Interventions: Behavioral: Family Integrated Care
- Family-Centered Care (FCC) (No Intervention): Infants assigned to usual FCC will have NICU nurses as primary caregivers per standard NICU protocol. FCC provides parents with orientation to the NICU; individualized teaching and support; and encouragement to participate in infant care under nursing supervision. Individualized support from social workers, lactation consultants and other specialists will be offered. As part of the study, parents will be asked to use the We3Health mobile app track their time in the NICU, time learning and time spent in infant caregiving activities and to keep of a journal of their NICU experience.

INTERVENTIONS:
Behavioral: Family Integrated Care — Parents of infants assigned to mFI-Care will be trained and treated as primary caregivers for their infants and participate in daily medical rounds, with mFI-Care-trained nurses serving as teachers and coaches.
  Arms: Family Integrated Care (mFI-Care)

SUMMARY:
The purpose of this study is to compare the standard of care in the neonatal intensive care unit (NICU), known as Family Centered Care, to a new model of care, called mobile enhanced Family Integrated Care. This exploratory two-group comparison study will examine the feasibility, acceptability and effectiveness, providing the first United States (US) information about outcomes of a new NICU care model that better integrates parents into all aspects of their baby's care. The use of mobile technology as part of this new model of care could improve access and equity in family integration for the many US families who face barriers to NICU involvement.

DETAILED DESCRIPTION:
Poor growth during neonatal intensive care unit (NICU) hospitalization is a modifiable risk factor contributing to mortality and serious long-term morbidity for many of the nearly 400,000 preterm infants born each year in the United States (US). Active parent involvement in preterm infant caregiving promotes parent-infant attachment and leads to higher breastfeeding rates, earlier discharge, and improved long-term neurodevelopment. Despite decades of evidence of the positive effects of parental involvement, parents remain for the most part passive bystanders in the NICU setting. Even with many NICUs adopting a Family-Centered Care (FCC) approach, parent-infant contact and parenting skills remain well below desired levels.

Family Integrated Care (FI-Care) is a novel intervention that differs from FCC because it formally teaches and supports parents to be primary caregivers for their infants and restructures the relationship between parents and clinicians so that parents are fully integrated into the care team. There is strong evidence from a large, well-designed cluster randomized trial conducted in Canada and Australia that FI-Care improves infant growth and breastfeeding rates and reduces maternal stress. However, these findings cannot be generalized to US NICUs where parents face many barriers to involvement in their infant's NICU care. The research team has developed a secure, HIPAA-compliant, mobile application to capture high quality data about parent involvement in NICU caregiving and to deliver essential elements of the FI-Care program remotely. This mobile-enhanced FI-Care (mFI-Care) may improve involvement of parents who cannot be present in the NICU during daytime hours due to distance, employment or other responsibilities and family commitments. Increasing access and equity in family-integrated care may improve outcomes for US preterm infants.

This exploratory two-group, multi-site comparison study will compare usual FCC with mFI-Care on growth and clinical outcomes of preterm infants < 33 weeks gestational age, as well as the stress, competence and self-efficacy of their parents. The feasibility and acceptability of using mobile technology to gather data about parent involvement in the care of preterm infants receiving FCC or mFICare as well as of the mFI-Care intervention will be evaluated (Aim 1). The effect sizes for infant growth (primary outcome) and for secondary infant and parent outcomes at NICU discharge and three months after discharge will be estimated (Aim 2). This study will provide important new information on innovative approaches to increasing parent involvement in NICU infant caregiving, including the use of a novel mobile application. The findings will be used to develop a future US cluster-randomized trial of mFI-Care with the aim of improving outcomes for preterm infants and their parents.

ELIGIBILITY:
Inclusion Criteria:

* Infant ≤ 33 weeks and their parent or guardian

Exclusion Criteria:

* Infant has a life-threatening congenital anomaly, is unlikely to survive or is receiving palliative care
* Parent is not English literate
* Parent < 18 years of age
* Parent does not have access to hand-held computer (smartphone or tablet)

Max Age: 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 347 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Change in infant weight (z-score) | 21 days of age after enrollment
  Z-score will be calculated by obtaining weight in kilograms from medical record and compared between the mFICare and usual FCC groups

SECONDARY OUTCOMES:
Amount of human milk/formula supplementation | At study enrollment and at hospital discharge, usually 21 days after admission
  number of ml for all breast feeding, breast pumping, bottle feeding, and nasal gastric (NG) feeding will be obtained from the medical record
Frequency of breastfeeding | At study enrollment and at hospital discharge, usually 21 days after admission
  Number of feedings for breast feeding, breast pumping, bottle feeding, and NG feeding will be obtained from the medical record
Breastfeeding rate | At study enrollment and at hospital discharge, usually 21 days after admission
  Breastfeeding rate will be calculated using amount of Number of feedings and ml for breast feeding, breast pumping, bottle feeding, and NG feeding will be obtained from the medical record
Length of stay | Number of days of NICU and hospital stay, usually 21 days after admission
  Number of days of NICU and hospital stay
Weight gain velocity | at NICU discharge, usually 21 days after admission
  number of grams gained from enrollment to specified date divided by the number of days = weight gain velocity
Major morbidities | at NICU discharge, usually 21 days after admission
  Nosocomial infection, necrotizing enterocolitis, intraventricular hemorrhage, retinopathy of prematurity, and adverse events.
Parent perceived stress | at NICU discharge, usually 21 days after admission
  Self- reported survey
Parenting competence | at NICU discharge, usually 21 days after admission
  self reported survey
Perceived parenting self-efficacy | at NICU discharge, usually 21 days after admission
  self-reported survey

OTHER OUTCOMES:
Change in infant weight (z-score) | 3 months post-discharge
  Z-score will be calculated by obtaining weight in kilograms from medical record and compared between the mFICare and usual FCC groups
Breastfeeding rate | 3 months post-discharge
  self-reported survey
Breastfeeding frequency | 3 months post-discharge
  self-reported survey
Hospital readmission rate | 3 months post-discharge
  self-reported survey
Perceived parenting self-efficacy | 3 months post-discharge
  self-reported survey

CONTACTS AND LOCATIONS:
Overall Officials: Linda Franck, RN, PhD, Principal Investigator — Dept of Family Care Nursing, California Preterm Birth Initiative, UCSF
Locations (6):
- United States (6):
  - Community Regional Medical Center, Fresno, California
  - Jacobs Medical Center, UC San Diego Health, La Jolla, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - UCSF Benioff Children's Hospital San Francisco, San Francisco, California
  - Kaiser Permanente - Santa Clara, Santa Clara, California
  - UCLA Medical Center, Santa Monica, Santa Monica, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Brien K, Bracht M, Robson K, Ye XY, Mirea L, Cruz M, Ng E, Monterrosa L, Soraisham A, Alvaro R, Narvey M, Da Silva O, Lui K, Tarnow-Mordi W, Lee SK. Evaluation of the Family Integrated Care model of neonatal intensive care: a cluster randomized controlled trial in Canada and Australia. BMC Pediatr. 2015 Dec 15;15:210. doi: 10.1186/s12887-015-0527-0. PMID 26671340
- [Derived] Franck LS, Magana J, Bisgaard R, Lothe B, Sun Y, Morton CH. Mobile-enhanced Family Integrated Care for preterm infants: A qualitative study of parents' views. PEC Innov. 2024 Apr 30;4:100284. doi: 10.1016/j.pecinn.2024.100284. eCollection 2024 Dec. PMID 38737891
- [Derived] Franck LS, Gay CL, Hoffmann TJ, Kriz RM, Bisgaard R, Cormier DM, Joe P, Lothe B, Sun Y. Neonatal outcomes from a quasi-experimental clinical trial of Family Integrated Care versus Family-Centered Care for preterm infants in U.S. NICUs. BMC Pediatr. 2022 Nov 22;22(1):674. doi: 10.1186/s12887-022-03732-1. PMID 36418988
- [Derived] Furtak SL, Gay CL, Kriz RM, Bisgaard R, Bolick SC, Lothe B, Cormier DM, Joe P, Sasinski JK, Kim JH, Lin CK, Sun Y, Franck LS. What parents want to know about caring for their preterm infant: A longitudinal descriptive study. Patient Educ Couns. 2021 Nov;104(11):2732-2739. doi: 10.1016/j.pec.2021.04.011. Epub 2021 Apr 17. PMID 33966954
- [Derived] Franck LS, Kriz RM, Bisgaard R, Cormier DM, Joe P, Miller PS, Kim JH, Lin C, Sun Y. Comparison of family centered care with family integrated care and mobile technology (mFICare) on preterm infant and family outcomes: a multi-site quasi-experimental clinical trial protocol. BMC Pediatr. 2019 Dec 2;19(1):469. doi: 10.1186/s12887-019-1838-3. PMID 31791285

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-17): https://cdn.clinicaltrials.gov/large-docs/70/NCT03418870/Prot_SAP_000.pdf